CLINICAL TRIAL: NCT04039360
Title: Self-expanding Metallic Stent Placement Followed by Neoadjuvant Chemotherapy and Scheduled Surgery for Treatment of Obstructing Left-sided Colonic Cancer
Brief Title: SEMS Placement Followed by Chemotherapy and Surgery for Obstructing Left-sided Colonic Cancer
Status: Completed | Type: Observational
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Zhen Jun Wang, Chairman of General Surgery, Beijing Chao Yang Hospital
Other Study IDs: SEMS-NCS-01
Record Dates: First submitted 2019-07-27; First posted 2019-07-31 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Complication of Treatment
Keywords: Left-sided colonic tumor; Intestinal obstruction; Self-expanding metallic stent; Neoadjuvant chemotherapy; Stoma
MeSH Terms: conditions — Intestinal Obstruction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: self-expanding metallic stent placement followed by neoadjuvant chemotherapy — Neoadjuvant chemotherapy was administered 1 week after successful SEMS placement and decompression for patient with obstructing left-sided colonic cancer. Patients received either three cycles of mFOLFOX6 repeated every 2 weeks or two cycles of CAPOX repeated every 3 weeks. Elective surgery was performed 2 weeks after completion of chemotherapy by experienced colorectal surgeons.

SUMMARY:
This study aimed to evaluate the safety and feasibility of SEMS followed by neoadjuvant chemotherapy prior to elective surgery for obstructing left-sided colon cancer.

DETAILED DESCRIPTION:
Stoma is reported to be frequent in self-expanding metallic stent (SEMS) treated patients with obstructing left-sided colon cancer than in those with non-obstructing surgery. Retrospective study reported worse overall survival with SEMS and elective surgery than with emergency surgery in patients with left-sided malignant colon obstruction. In practice, intestinal wall edema following stent placement increases the difficulty of surgery, and this could be a major problem if the interval between stent insertion and surgery is short (1-2 weeks). The patients with obstructing left-sided colon cancer received SEMS treatment, and the recevied neoadjuvant chemotherapy prior to elective surgery.

ELIGIBILITY:
Inclusion Criteria:

1. histologically proven adenocarcinoma located in the left colon (between the splenic flexure and 15 cm proximal to the anal margin)
2. Eastern Cooperative Oncology Group (ECOG) performance status of from 0 to 2

Exclusion Criteria:

1. history of any other cancer
2. multiple primary colorectal cancers
3. distant metastases
4. hereditary nonpolyposis colorectal cancer
5. familial adenomatous polyposis

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 11 patients included seven (63.6%) men and four (36.4%) women. The median age of the patients was 67 years (range, 43-72 years)
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2015-11-30 (Actual)

PRIMARY OUTCOMES:
stoma rate | 3 years after operation
  stoma rate after surgery

IPD SHARING:
Plan to Share IPD: Undecided